CLINICAL TRIAL: NCT01686698
Title: Study of the Effect of VSL#3 (Original De Simone Formulation) on Cognitive Function, Risk of Falls and Quality of Life in Patients With Cirrhosis
Brief Title: Effect of VSL#3 (Original De Simone Formulation) on Cognitive Function, Risk of Falls and Quality of Life in Patients With Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIBSP-VSL-2012-124
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Cirrhosis; Cognitive Dysfunction
Keywords: cirrhosis, VSL#3, cognitive function, falls, quality of life
MeSH Terms: conditions — Fibrosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL#3 (Original De Simone formulation) (Active Comparator): VSL#3 (Original De Simone formulation) sachets containing 450 x 109 bacteria, 1 sachet every 12 hours during 3 months (n=20).
  Interventions: Dietary Supplement: VSL#3 (Original De Simone formulation)
- Placebo (Placebo Comparator): Placebo sachets, 1 sachet every 12 hours during 3 months (n=20).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 (Original De Simone formulation) — VSL#3 (Original De Simone formulation) is a probiotic mixture of 8 proprietary strains, namely Streptococcus thermophilus, bifidobacteria and lactobacilli.
  Arms: VSL#3 (Original De Simone formulation)
Other: Placebo — Placebo will be formulated as identical in appearance and administered according to the same schedule as the active agent. Placebo contains maltose and silicon dioxide as inactive agent.
  Arms: Placebo

SUMMARY:
Probiotics, due to their ability to modulate intestinal flora, intestinal permeability and immune response, could decrease bacterial translocation and improve immune system alterations in cirrhosis. This could lead not only to improvement in liver function and to prevent bacterial infections and other complications but also to improve CD and to avoid its consequences falls, HRQoL deterioration).

Recently, the investigators have observed that VSL#3 administration to rats with experimental cirrhosis decreases bacterial translocation, inflammatory response and ascites formation, without changes in intestinal flora. This suggests an improvement in intestinal barrier that deserves further investigation.

VSL#3, through decreasing intestinal bacterial translocation and immune system modulation, could improve cognitive function and prevent the consequences of CD, including falls and HRQoL deterioration, in patients with cirrhosis.

DETAILED DESCRIPTION:
OBJECTIVES

Primary endpoint To assess the effect of VSL#3 on cognitive functions in patients with cirrhosis.

Secondary endpoint

To assess the effect of VSL#3 on:

* risk of falls
* HRQoL
* incidence of complications of cirrhosis and mortality during the study
* metabolomics in urine
* endocannabinoid system (MAGL and FAAH enzymes)
* soluble CD163 in blood as index of macrophage activation and portal hypertension (39)
* portal hypertension evaluated by abdominal doppler ultrasonography

PATIENTS AND METHODS

Inclusion criteria

Outpatients with cirrhosis cognitive dysfunction and/or falls in the previous year visited at Hospital de la Santa Creu i Sant Pau.

Cirrhosis will be diagnosed by clinical, analytical and ultrasonographic findings or by liver biopsy.

Exclusion criteria

* Hospitalization in the previous month due to decompensation of cirrhosis. Hepatocellular carcinoma or any other malignancy.
* Active alcohol intake (in the previous 3 months).
* Current overt acute or chronic hepatic encephalopathy.
* Clinically significant cognitive impairment according to Short Portable Mental Status Questionnaire (SPMSQ) > 5 points.
* Neurological disease.
* Inability to perform psychometric tests.
* Marked symptomatic comorbidities (cardiac, pulmonary, renal, untreated active depression).
* Life expectancy less than 6 months.
* Treatment with non-absorbable disaccharides.
* Treatment with antiviral drugs.
* Antibiotic treatment (norfloxacin).

Study Agent

VSL#3 is a probiotic mixture of 8 proprietary strains, namely Streptococcus thermophilus, bifidobacteria (B. breve, B. longum, B. infantis) and lactobacilli (L. paracasei, L. acidophilus, L. delbrueckii subsp bulgaricus, L. plantarum) . The active agent will be supplied as a 4.4g sachet at a dose of 450 billion live bacteria per sachet with maltose and silicon dioxide as excipients.

Placebo will be formulated as identical in appearance and administered according to the same schedule as the active agent. Placebo contains maltose and silicon dioxide as inactive agent.

VSL#3 is a food supplement which has been marketed in Europe since 2002. The study agent needs to be kept refrigerated at all times. It may be kept at room temperature for up to a week without affecting its potency.

Study agent will be supplied by Actial Farmaceutica Lda, Funchal (Portugal)

Study design

Double-blind placebo-controlled clinical trial.

Forty consecutive patients with cirrhosis and CD (PHES<-4) and/or falls in the previous year will be randomized to receive VSL#3, sachets containing 450 x 109 bacteria, 1 sachet every 12 hours during 3 months (n=20), or placebo (n=20).

Patients will be randomly assigned either to the active study agent or to the placebo and randomization list will be elaborated by a specific software and supplied by Actial Farmaceutica Lda.

The first box with the product (60 sachets) will be given to the patients at the beginning of the study. Patients will be instructed to take all the doses, to register if they miss some dose and to bring back the boxes at the next visit.

Patients will also be instructed to bring the urine samples in Falcon tubes that will be provided in the previous visit.

Then, the patients will give back the boxes and receive the next set of product every month. The investigators will count the number of remaining sachets in the returned boxes.

Patients will be visited at 0, 4, 6, 8, 12 and 20 weeks.

ASSESSMENTS

Patients will be visited at 0, 4, 6, 8, 12 and 20 weeks. The following patients' assessments will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with cirrhosis visited at Hospital de la Santa Creu i Sant Pau. Cirrhosis will be diagnosed by clinical, analytical and ultrasonographic findings or by liver biopsy.

Exclusion Criteria:

* Hospitalization in the previous month due to decompensation of cirrhosis. Hepatocellular carcinoma or any other malignancy.
* Active alcohol intake (in the previous 3 months).
* Current overt acute or chronic hepatic encephalopathy.
* Clinically significant cognitive impairment according to Short Portable Mental Status Questionnaire (SPMSQ) > 5 points.
* Neurological disease.
* Inability to perform psychometric tests.
* Marked symptomatic comorbidities (cardiac, pulmonary, renal, untreated active depression).
* Life expectancy less than 6 months.
* Treatment with non-absorbable disaccharides.
* Treatment with antiviral drugs.
* Antibiotic treatment (norfloxacin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
To assess the effect of VSL#3 (Original De Simone formulation) on cognitive function in patients with cirrhosis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: German Soriano, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain